CLINICAL TRIAL: NCT06423482
Title: Digitization Accuracy and Scannability of Two Different Implant-Supported Prosthodontic Framework Materials
Brief Title: Accuracy and Scannability of Implant-Supported Framework Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan Samy (Other)
Responsible Party: Sponsor-Investigator, Nourhan Samy, Ph.D student, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0796-11/2023
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Digitalization Accuracy
Keywords: Digitization; Accuracy; Trueness; Precision; Scannability; Implant-supported frameworks; Superstructures; Marginal adaptation; Titanium; PEEK

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEEK bar (Experimental)
  Interventions: Other: PEEK bar
- Titanium bar (Experimental)
  Interventions: Other: Titanium bar

INTERVENTIONS:
Other: PEEK bar — The framework will be constructed from Poly-Ether-Ether-Ketone (PEEK). The framework will be digitized by using a desktop scanner (Tabletop Scanner, Medit T-310; Medit Corp). The STL file produced will be considered as a reference file. Each framework will be scanned intraorally (n=10) by using an intraoral scanner (IOS) (Medit i700; Medit Corp).
  Arms: PEEK bar
Other: Titanium bar — The framework will be constructed from titanium. The framework will be digitized by using a desktop scanner (Tabletop Scanner, Medit T-310; Medit Corp). The STL file produced will be considered as a reference file. Each framework will be scanned intraorally (n=10) by using an intraoral scanner (IOS) (Medit i700; Medit Corp).
  Arms: Titanium bar

SUMMARY:
The present study aims to clinically evaluate and compare the scanning accuracy and the scannability of 2 different materials used in constructing frameworks for implant-supported prosthesis (titanium and PEEK).

The objective of the present study is to evaluate the digitization accuracy and scannability of milled titanium and PEEK implant-supported frameworks in intra-oral conditions and to evaluate the accuracy of the superstructures designed and constructed over the intraorally scanned framework.

DETAILED DESCRIPTION:
Background: For implementing a fully digital workflow, intraoral scanning of prosthetic frameworks may be required for editing purposes in some clinical scenarios. Different materials can be used in constructing implant-supported prosthetic frameworks. However, the scannability and the influence of the material used on the accuracy of the intraoral scan are still unclear.

Aim of the study: The purpose of this in vivo study is to evaluate the scanning accuracy and the scannability of different framework materials and to assess the marginal adaptation and accuracy of the superstructures designed and constructed over different scanned framework materials.

Materials and methods: Two milled maxillary implant-supported frameworks constructed from 2 different materials will be used in this study. Group I will be constructed from titanium and group II from Poly-Ether-Ether-Ketone (PEEK). The frameworks will be digitized by using a desktop scanner (Tabletop Scanner, Medit T-310; Medit Corp). The STL file produced will be considered as a reference file. Each framework will be scanned intraorally (n=10) by using an intraoral scanner (IOS) (Medit i700; Medit Corp). The STL files obtained from the intraoral scanner will be compared to the reference STL file to assess the scannability. The unscanned surface area in a preset time limit will be used to determine the scannability of each framework. To evaluate the scanning accuracy, all STL files will be imported into a surface-matching software program (Medit Design v3.0.6 Build 286; Medit Corp) where deviation measurements in (μm) will be calculated. A total of 20 superstructures made of nano-ceramic hybrid resin (Flexcera™ Smile Ultra) will be 3D-printed from each STL file obtained from intraoral scanning of the frameworks and then the marginal adaptation will be evaluated by using a stereomicroscope (SZ1145TR; Olympus, Japan). The accuracy will also be assessed by using a surface-matching software program (Geomagic Control X v.2018.1.1; 3D Systems).

Analysis: Data will be collected, tabulated, and statistically analyzed by using the appropriate statistical tests.

Keywords: Digitization, accuracy, trueness, precision, scannability, implant-supported frameworks, superstructures, marginal adaptation, titanium, PEEK, digital workflow, editing, nano-ceramic hybrid resin.

ELIGIBILITY:
Inclusion Criteria:

1. Maxillary edentulous adult patient with a good health status classified as ASA I or II physical status and having maxillary osseointegrated dental implants.
2. Adequate maxillary restorative space (6-8 mm).
3. Adequate zone of keratinized tissue (at least 2 mm).
4. Presence of an antagonistic dentate or rehabilitated arch.

Exclusion Criteria:

1. A systemic disease that compromises osseointegration such as uncontrolled diabetes mellitus or metabolic bone diseases.
2. Improper implant position.
3. Heavy smoking.
4. Inability to obtain written informed consent.

   -

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Digitization accuracy of the two different framework materials. | one year
  All scans obtained will be cropped eliminating soft tissue areas guided by the bar's finish line.
  The STL(D) file obtained from scanning the frameworks by using the desktop scanner will be used as reference scan for the assessment of trueness in the study, to measure the discrepancy with the corresponding 10 STLI files in each group.
  In each reference STL(D) file, the framework will be selected and used for alignment with their corresponding STL(I) with the best fit alignment algorithm to assess trueness, and then all the STL(I) in each material group will be superimposed to assess precision by using a specialized software program (Medit link). For the quantitative evaluation of 3D deviations between the reference STL(D) and the target data STL(I), the software program deviation display mode will be used to produce color-difference maps from which RMS (root mean square) will be calculated for statistical analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University, Alexandria, Stanly, Egypt

IPD SHARING:
Plan to Share IPD: Undecided